CLINICAL TRIAL: NCT06257238
Title: Virtual Reality For Shoulder Dysfunction Post Neck Dissection Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hayaa Khaled Yahya Aly, Physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004205
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: SHOULDER DYSFUNCTION
Keywords: SHOULDER DYSFUNCTION - NECK DISSECTION SURGERIES

STUDY DESIGN:
Intervention Model Description: Control group: (34 patients with shoulder dysfunction) receive traditional PT for shoulder dysfunction post neck dissection surgeries.
  Study group: (34 patients with shoulder dysfunction) receive fully immersive Head-Mounted Display virtual reality exercise plus traditional PT for shoulder dysfunction post neck dissection surgeries.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The study group includes 38 post neck dissection surgeries with shoulder dysfunction patients treated with fully immersive Head-Mounted Display virtual reality (Oculus Quest virtual reality (VR) headset with hand controller) for 30 min., each session includes three games exercise (Dance loop, Tennis and Boxing) with 10 min. for each game and 1 min. rest in between; in addition to their physical therapy program (Active ROM exercise for shoulder, Stretching exercise for shoulder extensors, adductors and internal rotators muscles and Strengthening exercise for shoulder muscles) 2 sessions per week for 2 months.
  Interventions: Device: Fully immersive Head-Mounted Display Virtual Reality; Behavioral: Traditional Physical Therapy Program
- Active comparator (Active Comparator): The study group includes 38 post neck dissection surgeries with shoulder dysfunction patients treated with traditional physical therapy program (Active ROM exercise for shoulder, Stretching exercise for shoulder extensors, adductors and internal rotators muscles and Strengthening exercise for shoulder muscles) 2 sessions per week for 2 months.
  Interventions: Behavioral: Traditional Physical Therapy Program

INTERVENTIONS:
Device: Fully immersive Head-Mounted Display Virtual Reality — patients are asked to wear the Oculus Quest VR on their heads and to hold the hand controllers by their hands and start the game exercises (Dance loop, Tennis ball and Boxing) with 10 min. for each game with 1 min. rest in between, plus the traditional PT program:(Active ROM exercise for shoulder, Stretching exercise for shoulder extensors, adductors and internal rotators muscles and Strengthening exercise for shoulder muscles) 2 sessions per week for 2 months.
  Other Names: Oculus Quest virtual reality headset with hand controller
  Arms: Experimental
Behavioral: Traditional Physical Therapy Program — patients are treated with Active ROM exercise for shoulder, Stretching exercise for shoulder extensors, adductors and internal rotators muscles and Strengthening exercise for shoulder muscles, 2 sessions per week for 2 months.

SUMMARY:
The goal of this clinical trial study: is to determine the effect of Virtual reality on pain and function for shoulder dysfunction post neck dissection surgeries. The main question is: Can Virtual reality technique affect the dysfunction of shoulder joint post neck dissection surgeries? Participants will receive the treatment for 2 times per week for 2 months. Assessment will be done before and after treatment.

DETAILED DESCRIPTION:
1. Subjects: sixty eight patients from both genders, suffering from shoulder dysfunction post neck dissection surgery, their ages ranges from 40-60 years.
2. Design of the study:

In this study the patients will be randomly assigned into two equal groups (34 patients for each group):

1. Group A (Study group):

   This group includes 34 patients suffering from pain and loss of shoulder flexion, abduction and external rotation ROM, patients will be treated with active ROM exercise, stretching exercise for shoulder extensors, adductors and internal rotators muscles and strengthening exercise for shoulder muscles, and with fully immersive Head-Mounted Display virtual reality (Oculus Quest virtual reality (VR) headset with hand controller) for 30 min. 2 times per week for 2 months.
2. Group B (Control group):

This group includes 34 patients suffering from pain and loss of shoulder flexion, abduction and external rotation ROM, patients will be treated with traditional physical therapy: active ROM exercise, stretching exercise for shoulder extensors, adductors and internal rotators muscles and strengthening exercise for shoulder muscles, 2 times per week for 2 months.

- Equipments:

Measuring tools:

* Measuring and assessment of pain by: Smart phone version of visual analogue scale (VAS).
* Measuring range of motion (ROM) by: Mobile application Goniometer.
* Measuring upper limb function by: The Arabic Version of Modified QuickDASH-9 Questionnaire.

Therapeutic equipment:

* Oculus Quest virtual reality (VR) headset with hand controller.

Each patient will play 3 games 10 min. for each with 1 min. rest in between. First game is Dance loop gameplay, there are throwing balls moving toward the patient in all directions, and the patient tries to catch all of them by the arm controllers, so it promote the movement of the arm toward flexion, abduction and external rotation directions.

Second game is Tennis ball, which promote the arm to move toward flexion, abduction and external rotation directions.

Third game is Boxing, which promote the arm to move toward flexion and abduction directions.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 40-60 years
* Both genders will participate in the study
* All patients have undergone neck dissection surgery
* All patients enrolled to the study will have their informed consent

Exclusion Criteria:

* Age more than 60 years or less than 40 years
* Subjects who have hearing problems
* Subjects who have visual problems
* Patients have acute viral diseases, acute tuberculosis, mental disorders or those with pace makers

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Smart phone version of visual analogue scale (VAS) | Assessing the change of the scores from baseline (beginning of treatment) to 2 months after treatment.
  Each patient determine his level of pain using an electronic version of a visual analogue scale, which is a validated, subjective measure for acute and chronic pain, by asking the user to mark a point on a line with minimum score of 0 "no pain" which is the best outcome and maximum score of 10 "worst pain possible" which is the worst outcome, which will be very helpful in the continuous monitoring of symptom diaries, feasible and efficient both for users and researcher.
Mobile application Goniometer | Assessing the change of the scores from baseline (beginning of treatment) to 2 months after treatment.
  One android mobile will be used in the study and the software will not be updated during data collection. Goniometer record apps will be used to measure shoulder range of movements (ROM)
The Arabic Version of Modified QuickDASH-9 Questionnaire | Assessing the change of The Arabic Version of Modified QuickDASH-9 Questionnaire score from baseline (beginning of treatment) to 2 months after treatment.
  The Arabic Modified Quick DASH-9, abbreviated from "Modified Quick Disabilities Arm Shoulder and Hand(DASH) questionnaire, is a single page; it consists of nine items extracted from The Quick DASH and DASH scales which concern the patient's upper extremity functions, with minimum score of 0 "no difficulty to perform all the activities" which is the best outcome and maximum score of 99 "unable to perform all the activities" which is the worst outcome.

CONTACTS AND LOCATIONS:
Overall Officials: H N Ashem, Professor, Study Director — faculty of physical therapy
Locations (1):
- Faculty of Physical Therapy, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feyzioglu O, Dincer S, Akan A, Algun ZC. Is Xbox 360 Kinect-based virtual reality training as effective as standard physiotherapy in patients undergoing breast cancer surgery? Support Care Cancer. 2020 Sep;28(9):4295-4303. doi: 10.1007/s00520-019-05287-x. Epub 2020 Jan 6. PMID 31907649
- [Background] El-Sayed D, Khalaf M, Hussein M. Psychometric properties of Arabic version of the modified QuickDASH-9 scale to measure the quality of recovery after dorsal hand burn injury. Int J Pharmtech Res. 2016;9(8):09-15.
- [Background] Patterson DR, Hoffman HG, Weichman SA, Jensen MP, Sharar SR. Optimizing control of pain from severe burns: a literature review. Am J Clin Hypn. 2004 Jul;47(1):43-54. doi: 10.1080/00029157.2004.10401474. No abstract available. PMID 15376608
- [Background] De Vet, H. C., Knol, D. L., Mokkink, L. B., and Terwee, C. B. (2011): Measurement in medicine: a practical guide. Cambridge university press.
- [Background] Mejia-Hernandez K, Chang A, Eardley-Harris N, Jaarsma R, Gill TK, McLean JM. Smartphone applications for the evaluation of pathologic shoulder range of motion and shoulder scores-a comparative study. JSES Open Access. 2018 Mar 13;2(1):109-114. doi: 10.1016/j.jses.2017.10.001. eCollection 2018 Mar. PMID 30675577
- [Background] Blough, D. K., Carrougher, G. J., Hoffman, H. G., Nakamura, D., Patterson, D. R. and Sharar, S. R. (2007)